CLINICAL TRIAL: NCT04420949
Title: High-precision Immersive Robotic Environment for Sensorimotor Training
Brief Title: Sensory Training for Visual Motion Sickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0632; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 5/1/2020 (Other: UW Madison); 1UL1TR002373-01 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-06-09 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Dizziness; Vertigo; Motion Sickness
Keywords: verticality; postural balance; visual dependence
MeSH Terms: conditions — Dizziness; Vertigo; Motion Sickness

STUDY DESIGN:
Intervention Model Description: The study will be conducted in three phases. The first phase is for baseline testing. The second phase is when treatment occurs. The third phase is for follow up testing. Participants will be tested twice during the baseline and follow up phases. Six treatment sessions will occur during the treatment phase.
Masking Description: It is not possible to mask this behavioral intervention. The study team small; thus, masking of the study team is also not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental): Healthy adults with visually-induced dizziness with undergo the testing and treatment.
  Interventions: Behavioral: Sensory re-weighting
- Vestibular-impaired (Experimental): Adults with unilateral or bilateral, peripheral vestibular loss who also have visually-induced dizziness with undergo the testing and treatment.
  Interventions: Behavioral: Sensory re-weighting

INTERVENTIONS:
Behavioral: Sensory re-weighting — During training, sensory re-weighting is driven by priming upregulation of somatosensory cues. Two rounds of training, each lasting 15 minutes and block-randomized in sets of 10 trials, are conducted per training visit. In each training trial, participants must determine the direction of gravity and then indicate if the rod being displayed is aligned with gravity or if it needs to rotate clockwise or counterclockwise for that to be so. Participants will be instructed to pay attention to what they feel from their feet, legs, and gut during training and to use that pressure, stretch, movement, and muscle tension feedback to help them sense gravity. Immediate auditory and non-orienting, visual feedback is provided after each trial. A staircase method is used to adapt the level of difficulty based on response accuracy. After two consecutive correct responses, the difficulty increases. After each incorrect response, the difficulty decreases. This process is repeated in each round.

SUMMARY:
This is a preliminary study to determine the reliability and validity of new tests of orientation and balance, as well as to test the effects of a new treatment for visually induced dizziness. Tests involve determining vertical alignment. The treatment is task-based and involves focusing attention on internal body sensations to help improve the sense of upright. Testing is done twice before and twice after treatment, which is provided twice-weekly during a three-week period between testing. The total time participants are involved in the study is approximately six weeks.

DETAILED DESCRIPTION:
Falls are a major concern for people living in countries all over the world. Tens of millions of people who fall are seriously injured and hundreds of thousands of people who fall die every year. People who are dizzy are far more likely to fall. The investigators are particularly interested in working with people who have dizziness that is caused by watching motion or looking at complex patterns (e.g. checkerboard patterns, walking through grocery store aisles, riding in vehicles, or watching movies).

This type of dizziness or vertigo is typically described as motion sickness or, more specifically, visually-induced dizziness. This problem affects adults who are healthy and adults who have a variety of health conditions. No diagnostic tests for this condition exist at this time and the treatments currently being used may result in worsening dizziness for some patients.

New tests were created for orientation and balance, as well as a new treatment for visually-induced dizziness. This is a preliminary study of the reliability and validity of the tests we developed, as well as whether the new treatment created results in reduced dizziness, improved balance, and changes in daily functioning.

It is not known whether the new tests of orientation and balance are better, worse, or the same as existing tests in the ability to detect problems, nor is it known if the new treatment technique is any better, worse, or the same as existing treatments for dizziness and imbalance. It is hypothesized that the new tests will be accurate and able to detect problems in impaired adults. Additionally, that the treatment will result in less dizziness, better balance, and reduced risk of falling.

The plan is to enroll a total of 30 people in this study, 15 who are healthy and 15 who have visually-induced dizziness due to a vestibular (inner ear) problem. Each participant will complete several questionnaires and tests of balance performance before and after undergoing the treatment. Participants attend 8 visits over 6 weeks. Each study visit lasts approximately 60 minutes.

During visits 1 and 2, which is a double baseline phase, the reliability and validity of the new testing procedures will be assessed. All participants will then enter the treatment phase (visits 2 through 7) and will attend twice-weekly appointments for three consecutive weeks. Following the treatment phase, participants will be re-assessed twice, immediately after (visit 7) and one week after (visit 8) completing treatment. During this phase, the short-term effectiveness of the treatment will be assessed.

Participants will complete questionnaires that measure the intensity of visually-induced dizziness, perceived handicap due to dizziness, and the impact of dizziness on daily functioning. Performance measures include the ability to determine what is upright based on the internal sense of gravity (verticality), standing upright, and walking-related balance tasks. The verticality tests are performed while the participant is secured in a harness and are either standing upright or tilted to the left or to the right. The testing task is to determine upright based on using internal body sensations. The standing balance test is performed on a platform that measures balance. The verticality tests and the standing balance test are experimental.

The treatment is task-based and is performed while the participant is supported in a harness and wearing virtual reality goggles. During the treatment, participants are either standing upright or tilted to the left or to the right. The treatment involves focusing attention on internal body sensations to help determine whether an image that is presented in an otherwise black virtual environment is aligned with gravity. Other visual and sound cues will be eliminated to prevent the use of these cues from influencing decisions about what is upright. As the participant becomes more successful at determining what is upright, the difficulty of the treatment task is gradually increased.

Participants symptoms will be monitored throughout the testing and treatment. Participants are given regular rest breaks and may request to rest at any time. Participation is voluntary and may be discontinued at any time.

The investigators anticipate only mild and infrequent side effects related to testing and treatment. The results of this study may influence how orientation and balance are assessed and how visually-induced dizziness is treated.

ELIGIBILITY:
Healthy Participants:

Inclusion Criteria: Participants must

* have normal self-reported cognitive function
* speak English fluently
* weigh less than 225 pounds and be less than 6'4"
* be able to support their body weight in an upright posture for 15 minutes at a time
* be able to follow the guidelines regarding permitted and prohibited additional treatments outlined in this protocol

Exclusion Criteria: Participants must not

* be pregnant or planning to become pregnant while in "on study" status
* have best-corrected visual acuity > 20/70
* have a self-reported, uncompensated, binocular vision abnormality, such as strabismus, amblyopia, or diplopia
* have peripheral neuropathy
* have a self-reported history of frequent syncope (>1/month)

Participants with Visually-induced Dizziness:

Inclusion Criteria: Participants must

* have self-reported symptoms of visually-induced dizziness
* have normal self-reported cognitive function
* speak English fluently
* weigh less than 225 pounds and be less than 6'4"
* be able to support their body weight in an upright posture for 15 minutes at a time
* be able to follow the guidelines regarding permitted and prohibited additional treatments outlined in this protocol

Exclusion Criteria: Participants must not

* be participating in vestibular and balance rehabilitation therapy and/or be pregnant or planning to become pregnant while in "on study" status
* have best-corrected visual acuity > 20/70
* have a self-reported, uncompensated, binocular vision abnormality, such as strabismus, amblyopia, or diplopia
* have peripheral neuropathy, and/or 5) have a self-reported history of frequent syncope (>1/month)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is not plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy | Vestibular-impaired
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy | Vestibular-impaired | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.02 (16.14) | 43.12 (16.78) | 42.07 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Visual Vertigo Analog Scale (VVAS) [Mean (Standard Deviation); unit: units on a scale] — The VVAS is a measure of the intensity of visual vertigo symptoms. The measure consists of a series of nine visual analog scales. Each scale ranges from 0 to 10. We report the total score, which is multiplied by 100. The range is from 0 to 900, and higher scores indicate greater severity of visual vertigo.
  units on a scale | 0 (0) | 163.4 (150.8) | 81.7 (132)

OUTCOME MEASURES:

1. Primary Outcome: Rod and Disk Test (RDT) Mean Performance
Description: An image of a rod will be shown in the central portion of the visual field. The surrounding virtual environment will be void. A batch of rod angles will be predetermined. This assessment will be completed using an Oculus Rift and without any reference to external visual cues. Only binocular testing will be completed. The average value for performance in each position will be used in data analysis. The mean of absolute value of the error in rod alignment measured in degrees for each body position tested will be used as the measurement variable for this outcome, and the primary outcome is the absolute value for mean performance in upright. In a prior study, the mean performance in this population is 0.39 (sd 0.8). Higher scores indicate subjective visual vertical alignment that is farther away from earth vertical.
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
degrees
  Visit 1 | 17 (7.5) | 13.3 (4)
  Visit 2 | 7.8 (8.8) | 12.1 (6.7)
  Visit 7 | 12.4 (6.7) | 10.3 (4.4)
  Visit 8 | 12.6 (5.3) | 10.3 (7)

2. Primary Outcome: Multisensory Balance Evaluation (MBE) as Measured by the Intersection Point Height
Description: This test is designed to assess balance during quiet standing in different sensory conditions. Participants perform one trial (lasting 30 seconds) of each condition. All trials are performed while standing on a force plate with the feet in a self-selected, comfortable position. The visual environment is controlled using an Oculus Rift. The surface conditions are either non-compliant or compliant. The frequency-dependent height of the Intersection Point (IP) of the ground reaction force is the main metric. The overall height of the IP curve obtained while the participant stands on a firm surface with their eyes open is the primary outcome. The height of IP ranges from 0 to 4.0, and higher values represent greater stability.
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
meters
  Visit 1 | 0.5 (0.23) | 0.53 (0.17)
  Visit 2 | 0.42 (0.18) | 0.52 (0.15)
  Visit 7 | 0.37 (0.17) | 0.39 (0.08)
  Visit 8 | 0.46 (0.15) | 0.37 (0.11)

3. Primary Outcome: Subjective Visual Vertical (SVV) Mean Performance
Description: as for outcome 1
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
degrees
  Visit 1 | -1.34 (1.65) | -1.3 (3.76)
  Visit 2 | -1.14 (1.36) | -1.4 (1.86)
  Visit 7 | -.21 (0.5) | -1.96 (1.17)
  Visit 8 | 1.0 (1.85) | -2.22 (2.08)

4. Primary Outcome: Rod and Frame Test (RFT) Mean Performance
Description: An image of a rod will be projected inside a tilted frame within the central portion of the visual field. The surrounding virtual environment will be void. The frame will be tilted by +/- 20° in the frontal plane. A batch of rod angles will be predetermined. This assessment will be completed using an Oculus Rift and without reference to external visual cues. Only binocular testing will be completed. The average value for performance in each position will be used in data analysis. The mean of absolute value of the error in rod alignment measured in degrees for each body position tested will be used as the measurement variable for this outcome, and the primary outcome is the absolute value for mean performance in upright. In a prior study, mean performance in this population is 6.51 (sd 7.8). Higher values indicate greater deviations of perceived vertical from earth vertical.
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
degrees
  Visit 1 | 3.9 (4.9) | 7.9 (2.9)
  Visit 2 | 5.7 (4.3) | 7.2 (3.3)
  Visit 7 | 5.6 (1.7) | 8.2 (6.1)
  Visit 8 | 7.6 (1.9) | 5.9 (3.45)

5. Secondary Outcome: Vision-related Dizziness Questionnaire (VRDQ) Total Score
Description: The VRDQ is used to quantify vision-related dizziness. This outcome measure consists of 25 questions comprising two subscales [frequency and severity of symptoms]. The range of scores for each sub-scale is 0 to 100 points. The total score is the average of both sub-scales. Higher scores represent greater frequency and severity of symptoms. Test-retest reliability for the VRDQ is well above the good performance level and convergent validity for the VRDQ was demonstrated with the Dizziness Handicap Inventory (DHI). Spearman correlation coefficients are 0.75 between the DHI and VRDQ frequency scale and 0.76 between the DHI and VRDQ severity scale.
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
units on a scale
  Visit 1 | 0 (0) | 90.8 (90)
  Visit 2 | 0 (0) | 86 (80)
  Visit 7 | 0 (0) | 74 (103)
  Visit 8 | 0 (0) | 76 (76)

6. Secondary Outcome: Dizziness Handicap Inventory (DHI) Total Score
Description: The DHI is used to assess the severity of self-perceived disability secondary to dizziness. The tool is comprised of 25 questions which are score as yes = 4 points, sometimes = 2 points, and no = 0 points. The total score has a range of 0 to 100 points. The reliability and validity of the DHI have been established.
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
units on a scale
  Visit 1 | 0.4 (0.9) | 19.2 (22)
  Visit 2 | 0.4 (0.9) | 24.4 (22.4)
  Visit 7 | 1 (2) | 23 (27)
  Visit 8 | 0.8 (1.1) | 18.4 (24.5)

7. Other Pre Specified Outcome: Activities-specific Balance Confidence Scale (ABCS) Average Score
Description: The ABCS is a measure of balance-related confidence. The scale is made up of 16 questions for which respondents rate their level of perceived confidence in not becoming unsteady or falling. The average score ranges from 0 to 100 percent. Higher scores indicate greater balance-related confidence. The reliability and validity of the ABCS has been established in adults with and without a history of falling.
Time Frame: Visit 1 (Week 1), Visit 2 (Week 2), Visit 7 (Week 4), and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
percent
  Visit 1 | 99 (0.8) | 91.8 (10)
  Visit 2 | 99 (1) | 88 (15)
  Visit 7 | 99 (1.3) | 93.5 (7.6)
  Visit 8 | 99 (0.7) | 95.6 (6.7)

8. Other Pre Specified Outcome: Vestibular Activities and Participation Measure (VAPM) Average Score
Description: The VAPM is a 34-item questionnaire that is used to assess the impact of vestibular dysfunction on daily activities and participation in various life roles. The psychometrics for this tool have been established for adults with vestibular disorders. The average score ranges from 0 to 4. Higher scores indicate greater impact of vestibular symptoms on daily activities and participation in various life roles.
Time Frame: Visit 1 (Week 1) and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
units on a scale
  Visit 1 | 0 (0) | 0.84 (0.79)
  Visit 8 | 0 (0) | 0.33 (0.48)

9. Other Pre Specified Outcome: Vestibular Rehabilitation Benefits Questionnaire (VRBQ) Total Score at the End of the Trial
Description: The VRBQ was developed to assess outcomes from vestibular rehabilitation. The 22 questions are based on a literature review, participant interviews, and items from other measures. These questions are divided into three sub-scales: dizziness and anxiety (6), motion provoked dizziness (5), and quality of life (11). The total score ranges from 0-100 percent and scores > 0 percent indicate the presence of symptoms, functional loss, or decreased quality of life. See http://www.isvr.soton.ac.uk/audiology/vrbq.htm for more information regarding the scoring methodology. It has been validated against other measures. The VRBQ is designed to measure the difference between the participant's current state of symptoms and quality of life compared to a state that is normal for the individual.
Time Frame: Visit 1 (Week 1) and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
percent
  Visit 1 | 5.4 (3.8) | 27.8 (27.7)
  Visit 8 | 2 (2.5) | 20.2 (28.4)

10. Other Pre Specified Outcome: Functional Gait Assessment (FGA) Total Score
Description: The FGA is a 10-item, observational, test of walking. Score for each item range from 0 to 3 and, thus, the total score ranges from 0 to 30. Use of an assistive device is permitted. Higher scores indicate greater stability during walking. The psychometrics of the FGA have been established for adults with balance disorders.
Time Frame: Visit 1 (Week 1) and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
units on a scale
  Visit 1 | 28.8 (1.6) | 29 (1.7)
  Visit 8 | 29.6 (0.89) | 29.3 (1.5)

11. Other Pre Specified Outcome: Walking Speed
Description: Gait speed has been shown to be a reliable and valid measure of functional balance in adults. Gait speed will be recorded during a 10-meter walk test. Participants will walk for 2-meters before entering and after exiting the 6-meter long recording section. A stopwatch will be used for timing.
Time Frame: Visit 1 (Week 1) and Visit 8 (Week 5)
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Healthy | Vestibular-impaired
Number analyzed (Participants) | 5 | 5
meters per second
  Visit 1 | 2.14 (0.20) | 2.05 (0.46)
  Visit 8 | 2.17 (0.27) | 2.17 (0.18)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Healthy | Vestibular-impaired
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Due to Covid-19 restrictions, enrollment in this study was lower than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04420949/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT04420949/ICF_000.pdf